CLINICAL TRIAL: NCT02674126
Title: When Are Parents Helpful? A Randomized Clinical Trial of the Efficacy of Maternal Sound for Pediatric Patients Undergoing Cardiac Surgery
Brief Title: The Efficacy of Maternal Sound for Pediatric Patients Undergoing Cardiac Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sayed Kaoud Abd-Elshafy, Associate Professor (Anesthesiology and Critical Care)- College of Medicine-Assiut University, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IRB000087350
Record Dates: First submitted 2016-01-31; First posted 2016-02-04 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Maternal-Fetal Relations
Keywords: Cardiac Surgery; Maternal sound; Cortisol; Blood sugar; Stress
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (Placebo Comparator): Control group
  Interventions: Behavioral: Control group
- Maternal sound group (Active Comparator): Maternal sound
  Interventions: Behavioral: Maternal sound group

INTERVENTIONS:
Behavioral: Control group — Patients in the control group listened to a blank CD connected to the patient ears before induction of anesthesia and continued during intra operative period till extubation in intensive care unit
  Arms: Control group
Behavioral: Maternal sound group — The recorded maternal voice (while they are singing the most popular songs their children like or telling a story to help their children to sleep) listened by CD player connected to the patient ears before induction of anesthesia and continued during intra operative period till extubation in intensive care unit
  Arms: Maternal sound group

SUMMARY:
A newborn's recognition and preference for their mother's voice occurs early in life, very likely during fetal development. Maternal voice stimuli undergo a unique form of cerebral processing that lends support for the existence of neurophysiologic mechanisms that reflect a child's preference for his/her mother's voice. This study aims to evaluate and compare the effect t of maternal sound listening in children undergoing cardiac surgery on stress response and physiological parameters.

DETAILED DESCRIPTION:
Children (4 to 8 years) undergoing repair of Atrial Septal Defect (ASD). Patients will be randomized into two equal groups (30 in each group) (control group and maternal sound group); in control group patients listened to a blank CD, while in maternal sound group patients listened to a recorded CD where the mother singing the most popular songs their children like or telling a story to their children. Baseline stress markers (blood glucose and plasma cortisol) sampled the morning before scheduled operation. A interview with the patients and their parents before operation to collect the questionnaire regarding patient's characteristic (age, sex, weight and height), patient's clinical data (medical diagnosis and American Society of Anesthesiologists physical status) and haemodynamic data (blood pressure, heart rate, oxygen saturation on room air, temperature). In addition, the researcher interviewed with the mothers to record on one CD their voice while they are singing the most popular songs their children like or telling a story to their children to help them to sleep to be used during intra-operative period in maternal sound group.

ELIGIBILITY:
Inclusion Criteria:

* Age range 4-8 years
* Elective cardiac surgery
* Atrial Septal Defect (ASD) repair with Cardiopulmonary bypass

Exclusion Criteria:

* Previous cardiac surgery
* Diabetes mellitus
* Hearing impairment
* Psychiatric illness
* Neurological illness.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 106 (Actual)
Dates: Start 2016-01; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Blood cortisol level | Up to 24 hours
  Blood sample will be taken at preoperative, at sternotomy, after 10 minutes of cross clamping during cardiopulmonary bypass, during rewarming and at extubation
Blood sugar level | Up to 24 hours
  Blood sample will be taken at preoperative, at sternotomy, after 10 minutes of cross clamping during cardiopulmonary bypass, during rewarming and at extubation

SECONDARY OUTCOMES:
Pain assessment | Within the first 24 hours
  Pain assessment after extubation by Objective Pain Scale (OPS)
Sedation assessment | Within the first 24 hours
  Sedation assessment after extubation by Richmond Agitation Sedation Scale (RASS)
Post Traumatic Stress Disorder | Within the first postoperative week
  An interview conducted with the patients and their parents by researcher blinded to the group randomization within the first postoperative week
Post hospital behavior questionnaire | Within the first postoperative week
  An interview conducted with the patients and their parents by researcher blinded to the group randomization within the first postoperative week

CONTACTS AND LOCATIONS:
Overall Officials: sayed abd elshafy, Principal Investigator — associate professor
Locations (1):
- Faculty of Medicine, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided